CLINICAL TRIAL: NCT04496544
Title: Safety Assessment of Femoropopliteal Endovascular Treatment With PAclitaxel-coated Devices (SAFE-PAD Study)
Acronym: SAFE-PAD
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Medtronic (Industry); Philips Healthcare (Industry); Bard Peripheral Vascular, Inc. (Industry); Boston Scientific Corporation (Industry); Cook Medical (Unknown)
Responsible Party: Principal Investigator, Eric Secemsky, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2019P000950
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Arterial Disease; Paclitaxel Adverse Reaction; Safety Issues
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Drug-Coated Devices: Medicare fee-for-service beneficiaries who underwent femoropopliteal artery revascularization with drug-coated devices (drug-eluting stent ± drug-coated balloon, bare metal stent with drug-coated balloon, or drug-coated balloon alone)
  Interventions: Other: Retrospective data collection
- Non-Drug-Coated Devices: Medicare fee-for-service beneficiaries who underwent femoropopliteal artery revascularization with non-drug-coated devices (bare metal stent ± percutaneous transluminal balloon angioplasty or percutaneous transluminal balloon angioplasty alone)
  Interventions: Other: Retrospective data collection

INTERVENTIONS:
Other: Retrospective data collection — No intervention; retrospective data collection

SUMMARY:
The SAFE-PAD Study aims to evaluate the long-term safety of paclitaxel-coated devices compared with non-paclitaxel-coated devices for femoropopliteal artery revascularization among a broad, real-world population of patients with peripheral artery disease. This multi-year analysis aims to create an ongoing mechanism to evaluate the safety of paclitaxel-coated devices in real world practice. The null hypothesis is that the paclitaxel-coated devices are associated with an increase in mortality relative to the non-drug-coated devices beyond an acceptable magnitude (i.e. the non-inferiority margin), and the alternative hypothesis is that paclitaxel-coated devices are not associated with an increase in mortality relative to the non-drug-coated devices beyond the non-inferiority margin.

DETAILED DESCRIPTION:
This is an observational retrospective cohort study using claims data to evaluate the long-term safety of paclitaxel-coated devices compared with non-drug coated devices for femoropopliteal artery revascularization, with median follow-up time for the population surpassing 5 years. A series of supplemental sensitivity analyses will be conducted to assess and mitigate the potential for unmeasured confounding and to determine the impact of repeat interventions and paclitaxel exposure on survival. Finally, sub-group analyses will be performed to investigate whether there is differential safety of paclitaxel-coated devices across different patient profiles.

ELIGIBILITY:
Inclusion Criteria:

* All fee-for-service Medicare beneficiaries who underwent femoropopliteal artery revascularization. Patients are allowed to undergo simultaneous revascularization of lesions outside this target vessel during the same procedure.
* All patients with ≥1 year of Medicare claims data prior to their index procedure.

Exclusion Criteria:

* Patients without 1 year of Medicare claims data prior to their index revascularization procedure.
* Patients that do not have both a carrier file charge and an institutional file charge on the date of an outpatient procedure. This removes procedures performed in certain clinical settings, such as office-based clinics, that do not submit the Healthcare Common Procedure Coding System (HCPCS) code needed to identify drug-coated devices.

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study cohort will include all Medicare fee-for-service beneficiaries who underwent femoropopliteal artery revascularization with either drug-coated devices (drug-eluting stent [DES] ± drug-coated balloon [DCB], bare metal stent [BMS] with DCB, or DCB alone) or non-drug-coated devices (BMS ± percutaneous transluminal angioplasty [PTA] or PTA alone). Each group will additionally be composed of two device-specific subgroups: a DCB sub-group and DES sub-group in the drug-coated group, and a PTA sub-group and a BMS sub-group in the non-drug group.
Sampling Method: Non-Probability Sample
Enrollment: 168553 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Time from index procedure date to the date of death, to be updated periodically until the median duration of follow-up for the cohort reaches 5 years
  All-cause mortality of patients who underwent femoropopliteal artery revascularization with drug-coated devices or non-drug-coated devices

SECONDARY OUTCOMES:
Repeat hospitalization | 1, 2 and 3 years after index procedure
  Rates of repeat hospitalization
Repeat endovascular or surgical revascularization | 1, 2 and 3 years after index procedure
  Rates of repeat endovascular or surgical revascularization
Target vessel revascularization | 1, 2 and 3 years after index procedure
  Rates of target vessel revascularization among inpatient procedures
Lower extremity amputation | 1, 2 and 3 years after index procedure
  Rates of lower extremity amputation
Optimal medical therapy | 1, 2 and 3 years after index procedure
  Rates of optimal medical therapy

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Secemsky, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Robert W Yeh, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
As restricted by the data use agreement with the Centers for Medicare and Medicaid Services (CMS), we will not allow any data sharing for this project and we will not make any distribution of the CMS data.

REFERENCES:
- [Derived] Secemsky EA, Song Y, Schermerhorn M, Yeh RW. Update From the Longitudinal Assessment of Safety of Femoropopliteal Endovascular Treatment With Paclitaxel-Coated Devices Among Medicare Beneficiaries: The SAFE-PAD Study. Circ Cardiovasc Interv. 2022 Jun;15(6):e012074. doi: 10.1161/CIRCINTERVENTIONS.122.012074. Epub 2022 May 20. No abstract available. PMID 35593638
- [Derived] Secemsky EA, Raja A, Shen C, Valsdottir LR, Schermerhorn M, Yeh RW; SAFE-PAD Investigators. Rationale and Design of the SAFE-PAD Study. Circ Cardiovasc Qual Outcomes. 2021 Jan;14(1):e007040. doi: 10.1161/CIRCOUTCOMES.120.007040. Epub 2021 Jan 13. PMID 33435732